CLINICAL TRIAL: NCT00651898
Title: Comparison of a Circulating-water Garment With a Combination of Forced-air Warming and Circulating-water Mattress Warming During Major Abdominal Surgery
Brief Title: Circulating-water Garment With Forced-air Warming and Circulating-water Mattress During Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, d sessler, MD, The Cleveland Clinic
Other Study IDs: 06-597
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Hypothermia
Keywords: abdominal surgery; hypothermia; circulating water mattress
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: This group will receive the circulating water garment
- B: This group will receive the circulating water mattress and be covered by a forced air warming device for both the upper body and lower body connected to two warmers.

SUMMARY:
The purpose of this study is to see if the combination of a circulating water mattress beneath the patient combined with forced air warming over top of the patient will prevent hypothermia (low body temperature) just as well as a garment that circulates warm water around the patient, during your major abdominal surgery. Patients will be randomly assigned to one of these two groups.

DETAILED DESCRIPTION:
Group A: This group will receive the circulating water garment Group B: This group will receive the circulating water mattress and be covered by a forced air warming device for both the upper body and lower body

Once the patient is moved to the operating room table, the surface of the back will begin to be warmed using either the circulating-water garment for those in Group A or the circulating-water mattress for those in Group B. Following the start of anesthesia, additional warming will be done by covering the large parts of the legs and the upper and side of the chest using either the circulating-water garment for those in Group A or upper- and lower-body forced-air warmers for those in Group B.

Patient involvement will last until the warming devices are removed prior to departure from the operating room. There is no follow-up to this study.

ELIGIBILITY:
Inclusion Criteria:

* MaJor abdominal surgery
* Age between 18 and 85 years.

Exclusion Criteria:

* Fever (core temperature >38°C)
* Combined procedures (e.g.: simultaneous liver and kidney transplantation)
* Contraindication to forced-air or circulating-water warming which would be impacted by use of warming blanket
* Anticipated veno-venous bypass
* Current Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients between 18-85 years of age who are undergoing major abdominal surgery who do not have a contradiction to forced-air or circulating water warming. Patient's undergoing combined procedures are not eligible to participate. Patient can not have a core temperature over 38°C, be pregnant or
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2006-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome will comprise the difference between the pre-induction temperature and the intraoperative temperature | Every 15 minutes throughout surgery

CONTACTS AND LOCATIONS:
Overall Officials: Maged Argalious, MD, Principal Investigator — The Cleveland Clinic; Daniel I Sessler, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perez-Protto S, Sessler DI, Reynolds LF, Bakri MH, Mascha E, Cywinski J, Parker B, Argalious M. Circulating-water garment or the combination of a circulating-water mattress and forced-air cover to maintain core temperature during major upper-abdominal surgery. Br J Anaesth. 2010 Oct;105(4):466-70. doi: 10.1093/bja/aeq170. Epub 2010 Aug 3. PMID 20685683